CLINICAL TRIAL: NCT07233837
Title: Hydrogen Peroxide and Ultraviolet Light for Disinfecting Surfaces in Intensive Care Units: A Randomized, Controlled, Cluster, Crossover Clinical Trial
Brief Title: Hydrogen Peroxide and Ultraviolet Light for Disinfecting Surfaces in Intensive Care Units
Acronym: Hylight
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Hospital Sírio-Libânes, São Paulo, Brazil (Unknown); Hospital do Coracao (Other); Beneficência Portuguesa de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CAAE 71265723.0.1001.0071
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Infection, Hospital; Antimicrobial; Pneumonia Associated With Mechanical Ventilation; Urinary Tract Infection(UTI); Catheter Related Blood Stream Infections
Keywords: Healthcare associated infections; Antimicrobial use; Intensive care units; pneumonia, ventilator-associated; Catheter-related infections; Urinary tract infections; Hydrogen Peroxide; Ultraviolet light
MeSH Terms: conditions — Cross Infection; Urinary Tract Infections; Pneumonia, Ventilator-Associated; Catheter-Related Infections | interventions — Hydrogen Peroxide; Ultraviolet Rays

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, cluster, crossover, trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Surface disinfection with aerosolized hydrogen peroxide (Experimental): The hygiene team of each participating ICU will spray aerosolized peroxide hydrogen using a specific device when performing terminal cleaning of the ICU bed after the patient's discharge. As peroxide hydrogen aerosol can be irritating to people nearby, we will use a tent designed to cover the bed and nearby equipment during peroxide hydrogen disinfection, thus preventing aerosols from spreading to other beds and other areas of ICUs where beds are not in closed rooms.
  Interventions: Other: Aerosol of hydrogen peroxide
- Surface disinfection with irradiation of ultraviolet light (Experimental): The hygiene team of each participating ICU will use a specific device, requiring no manipulation, for irradiating UV light for the purpose of disinfecting beds and surfaces near beds during terminal cleaning. To prevent UV irradiation from reaching occupied beds and other areas of the ICU, the same tent described in the "peroxide hydrogen" arm.
  Interventions: Other: Irradiation of ultraviolet light
- Usual disinfection (No Intervention): The control group will perform standard cleaning and disinfection of the beds and the environment according to their previous protocols, using the usual products.

INTERVENTIONS:
Other: Aerosol of hydrogen peroxide — Spray of aerosolized peroxide hydrogen using a specific device when performing terminal cleaning of the ICU bed after the patient's discharge.
  Other Names: Hydrogen Peroxide
  Arms: Surface disinfection with aerosolized hydrogen peroxide
Other: Irradiation of ultraviolet light — Irradiation of UV light for the purpose of disinfecting beds and surfaces near beds during terminal cleaning.
  Other Names: Ultraviolet light
  Arms: Surface disinfection with irradiation of ultraviolet light

SUMMARY:
Healthcare-associated infections (HAIs) remain a major problem in intensive care units (ICUs), driven by environmental contamination with multidrug-resistant organisms that persist despite routine manual cleaning. While hydrogen peroxide aerosolization and ultraviolet-C light devices have shown promise in reducing surface contamination, current evidence is inconsistent, mostly derived from single-center studies, and rarely linked to patient-centered outcomes.

The investigators will conduct this cluster-randomized, crossover trial in 12 Brazilian ICUs. Each ICU will sequentially implement three strategies: (1) usual surface disinfection; (2) usual surface disinfection followed by hydrogen peroxide aerosolization at 7.9% concentration, applied through a dedicated device inside a protective tent during terminal cleaning of patient beds; and (3) usual surface disinfection followed by automated ultraviolet-C irradiation, also applied under the same tent to shield adjacent occupied beds.

The primary outcome will be the average duration of antimicrobial therapy, with secondary outcomes including HAI incidence, environmental contamination with multidrug-resistant organisms, specific HAIs (associated-ventilator pneumonia, central-line associated bloodstream infection, and catheter-associated urinary tract infection), and ICU length of stay costs.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years and older who will be admitted to the participating ICUs

Exclusion Criteria:

* Patients under 18 years
* ICUs that use peroxide hydrogen or ultraviolet light for surface disinfection as part of their protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4800 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2027-02-26 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Duration of antimicrobial therapy | 3 months
  Number of days each included patient used antimicrobial therapy during ICU admission

SECONDARY OUTCOMES:
Healthcare-associated infections | 3 months
  Density of healthcare-associated infections during ICU admission
Contamination of environmental surfaces by multi-resistant microorganisms | 3 months
  We will collect environmental samples from 4 surfaces highly touched by the patient, health team and family (bed rails, monitor and infusion pump buttons, meal table or procedure table, and IV drip stand) before and after the intervention. For analysis of the environmental samples, characterization of the density and microbiological profile of biofilms on the different surfaces of the ICU beds will be performed using large-scale DNA sequencing techniques associated with bioinformatics analysis.
Incidence density of ventilator-associated pneumonia | 3 months
Incidence density of central line-associated bloodstream infections | 3 months
Incidence density of catheter-associated urinary tract infection | 3 months
Intensive care unit length of stay costs | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio P Nassar Jr, PhD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (12):
- Brazil (12):
  - Hospital Maternidade Sao Vicente De Paulo, Barbalha, Ceará
  - Instituto Hospital de Base, Brasília, Federal District
  - Hospital Estadual de Aparecida de Goiânia, Aparecida de Goiânia, Goiás
  - Santa Casa de Misericórdia de Passos, Passos, Minas Gerais
  - Fundo Municipal de Saúde de Maringá, Maringá, Paraná
  - Hospital da Restauração, Recife, Pernambuco
  - Hospital Universitário da Universidade Federal do Piauí, Teresina, Piauí
  - Hospital Universitário Onofre Lopes, Natal, Rio Grande do Norte
  - Hospital Geral de Caxias do Sul, Caxias do Sul, Rio Grande do Sul
  - Hospital de Pronto Socorro de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Dr Leo Orsi Bernardes, Itapetininga, São Paulo
  - Hospital Pelópidas Silveira, Recife

IPD SHARING:
Plan to Share IPD: No
The sharing of individual participant data is subject to approval by the Institutional Review Boards and the Brazilian Ministry of Health.